CLINICAL TRIAL: NCT04955652
Title: Evaluation of Best Practice Alerts and an Actionable Sidebar in Electronic Health Records in Promoting Bone Densitometry Scans
Brief Title: Evaluation of Alerts in Promoting Bone Densitometry Scans
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: A conflicting project required the same sample for a different purpose.
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Amir Goren, Program Director, Behavioral Insights Team, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020-0996
Record Dates: First submitted 2021-06-22; First posted 2021-07-09 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Bone Diseases; Communication
Keywords: Bone Diseases; Alerts; Densitometry; Dual Energy X-ray Absorptiometry Scan
MeSH Terms: conditions — Bone Diseases; Communication

STUDY DESIGN:
Intervention Model Description: 1 x 2 factorial design, with randomization happening at the patient level
Who Masked: Participant, Care Provider
Masking Description: The participants and providers will not know that alerts were randomized. Participants will not know the arm to which they were assigned. Providers might notice that a given participant did or did not receive a certain alert, but this is expected to be unlikely, given the volume of alerts to which providers are exposed constantly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): A health maintenance topic, actionable sidebar item, and a single-click best practice alert are presented.
  Interventions: Behavioral: Health Maintenance Topic; Behavioral: Actionable Sidebar Item; Behavioral: Best Practice Alert
- Silent Best Practice Alert (Experimental): A health maintenance topic and an actionable sidebar item are presented. The best practice alert is set to be silent and will not appear in the patient's chart.
  Interventions: Behavioral: Health Maintenance Topic; Behavioral: Actionable Sidebar Item

INTERVENTIONS:
Behavioral: Health Maintenance Topic — Alert
  Other Names: HMT
Behavioral: Actionable Sidebar Item — Alert
  Other Names: Storyboard
Behavioral: Best Practice Alert — Alert
  Other Names: BPA
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to assess, prospectively, the effect of provider-facing alerts for bone densitometry scans with and without a single-click best practice alert (BPA) on scan orders and completions. The investigators hypothesize that the remaining alerts left in place (via health maintenance topics and an actionable item in the electronic health record sidebar) will be as effective without the BPA compared to the alerts with a BPA.

DETAILED DESCRIPTION:
Standard care for bone densitometry scans at Geisinger--i.e., dual-energy x-ray absorptiometry (DXA) scans--involves (1) an alert under the health maintenance topics tab in Epic, (2) an actionable item in a sidebar (Storyboard), (3) and a single-click best practice alert (BPA). Storyboard and the BPA theoretically serve a redundant function, but it is possible that combined alerting is effective. Therefore, the investigators plan to evaluate whether the BPA for DXA scans will increase the percentage of DXA scans ordered and completed.

For this evaluation, the investigators will randomly assign (by odd and even MRN) half of patients who need DXA scans to go through standard care (including the single-click BPA) and half of patients to have no BPA shown to their provider, but only the health maintenance topic and actionable Storyboard alert. This evaluation will help the investigators determine whether redundant, more traditional alerts such as BPAs are helpful or can be removed from alerts for DXA scans.

The randomization of patients to different alert conditions will be in place until 4,200 participants have been reached (estimated sample to detect 4% absolute difference, rounded to nearest hundred) or 6 months, whichever comes first. To account for delays in updating clinical databases, the outcome data will pulled 3 months after each encounter (for a maximum study period of 9 months).

The main analysis will use a logistic regression to compare the two groups. Exploratory analyses will also examine the time from order to completion to examine any effect on timing between arms. Another set of exploratory analyses will also examine the number of other BPAs firing to see if alert fatigue influenced the number of orders or completions or interacted with the experimental conditions.

ELIGIBILITY:
Inclusion Criteria:

* In primary care
* Records indicate patient is due for a bone densitometry scan (generally, a high-risk patient that requires this scan or age 65 and older)

Exclusion Criteria:

* Encounters at clinics/sites where the randomization build cannot easily be deployed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Bone Densitometry Scan Order Placed | 6 months or as long as it takes to reach N=4,200, whichever occurs first
  Binary variable indicating whether or not the order was placed

SECONDARY OUTCOMES:
Bone Densitometry Scan Completed | 6 months or as long as it takes to reach N=4,200, whichever occurs first
  Binary variable indicating whether or not the order placed at the encounter was completed

OTHER OUTCOMES:
Bone Densitometry Scan Completion Time | 6 months or as long as it takes to reach N=4,200, whichever occurs first
  Number of days from order time to completion time
Number of Unique Alerts | 6 months or as long as it takes to reach N=4,200, whichever occurs first
  Number of unique alerts (BPAs and medication alerts) that fired at the encounter
Number of Alerts Fired | 6 months or as long as it takes to reach N=4,200, whichever occurs first
  Number of alerts (BPAs and medication alerts) that fired at the encounter
Total number of BPAs | 6 months or as long as it takes to reach N=4,200, whichever occurs first
  Total number of BPAs that fired at the encounter
Total number of medication alerts | 6 months or as long as it takes to reach N=4,200, whichever occurs first
  Total number of medication alerts that fired at the encounter
Total number of passive alerts | 6 months or as long as it takes to reach N=4,200, whichever occurs first
  Total number of passive alerts that fired at the encounter
Total number of interruptive alerts | 6 months or as long as it takes to reach N=4,200, whichever occurs first
  Total number of interruptive alerts that fired at the encounter

CONTACTS AND LOCATIONS:
Overall Officials: Amir Goren, PhD, Principal Investigator — Program Director, Behavioral Insights Team

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency. This will include the essential data and code needed to replicate the analysis that yielded reported findings. The PI did not examine or analyze any data from this study prior to this registration.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The data will become available after publication of study results in a scientific journal and will be available as long as the Open Science Framework hosts the data.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.